CLINICAL TRIAL: NCT06236828
Title: The MRI-based Evaluation of Safety and Efficacy of EVT and SMT: A Retrospective, Multicenter Study
Status: Completed | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: MR-EPICS
Record Dates: First submitted 2023-11-29; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-01

CONDITIONS: Stroke; Acute Ischemic Stroke; Ischemic Stroke
Keywords: MRI; Endovascular Thrombectomy; Standard Medical Therapy; Large Vessel Occlusion; Acute Basilar Artery Occlusion
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endovascular Thrombectomy: For patients who onset within 4.5 hours and meet the criteria for intravenous thrombolysis treatment, they could receive intravenous thrombolysis treatment beforehand and bridging to endovascular therapy.
  Interventions: Device: Mechanical Thrombectomy
- Standard Medical Therapy: For patients who onset within 4.5 hours and met the criteria for intravenous thrombolysis treatment, recombinant tissue plasminogen activator (rt-PA) or urokinase, and other intravenous thrombolysis therapies should be pre-administrated.

INTERVENTIONS:
Device: Mechanical Thrombectomy — The endovascular mechanical thrombectomy methods mainly include stent retriever thrombectomy, ADAPT thrombus aspiration technique, or their combination.
  Groups: Endovascular Thrombectomy

SUMMARY:
Acute Basilar Artery Occlusion (ABAO), a condition with a high risk of mortality or disability (up to 80%). The safety and efficacy of endovascular thrombectomy (EVT) in ABAO remains uncertain due to inconsistent evidence from random controlled trials (RCTs).

Recent studies have explored the use of MRI in ABAO, this study aims to assess the efficacy and safety of EVT and standard medical therapy (SMT) in the treatment of ABAO within 24 hours of onset. It also aims to explore the feasibility and prognostic value of MRI-based assessment of ABAO infarction using AI image analysis software.

ELIGIBILITY:
Inclusion Criteria:

1. Preliminary diagnosis of posterior circulation ischemic stroke based on clinical symptoms or imaging examinations.
2. Confirmation through CTA/MRA/DSA that there is occlusion of the basilar artery or the V4 segment of the vertebral artery leading to functional occlusion of the basilar artery.
3. Age 18 years and older.
4. Symptom onset within 24 hours.
5. Having a baseline MRI evaluation, including at least DWI and T2 FLAIR sequences (baseline MRI for the EVT group before the operation; baseline MRI for the SMT group within the treatment window (within 4.5 hours of onset) for thrombolytic patients before or during the thrombolysis process should initiate as early as possible; baseline MRI for the SMT group for extended treatment window patients (between 4.5 hours to 12 hours of onset) should initiate as early as possible).

Exclusion Criteria:

1. mRS score ≥ 3 before onset;
2. Significant neuroimaging changes such as cerebral hemorrhage, cerebellar mass lesion, acute hydrocephalus, etc., are present;
3. Lack of follow-up results within 90 days after operation;
4. Life expectancy < 3 months;
5. Baseline imaging and crucial clinical data are missing;
6. Special cases involving pregnancy and lactation;
7. Severe systemic diseases or advanced cancer that may potentially interfere with the prognosis;
8. Allergic reactions to contrast agents or nickel-titanium alloys;
9. Currently participating in other clinical trials;
10. Pre-existing neurological disorders or psychiatric conditions that could affect the assessment of the disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2020 to September 2022, ABAO patients at Xuanwu Hospital Capital Medical University and 10 branch centers underwent EVT or SMT.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Rate of modified Rankin Scale (mRS) score of 0-3 at 90 days | 90 days after EVT or SMT
  The mRS score range from 0 (no disability) to 6 (death)

SECONDARY OUTCOMES:
Mortality | 90 days after EVT or SMT
  Death defined as a mRS score of 6
Rate of mRS score of 0-2 | 90 days after EVT or SMT
  The mRS score range from 0 (no disability) to 6 (death)
Improvement of mRS score | 90 days after EVT or SMT
  The mRS score range from 0 (no disability) to 6 (death)
  The mRS score range from 0 (no disability) to 6 (death)
Change of the National Institutes of Health Stroke Scale (NIHSS) score comparing to baseline | 24 hours and 5-7 days (or at discharge) after EVT
  The NIHSS score range from 0 (no deficit) to 42 (maximum deficit).
Rate of successful revascularization (mTICI 2b-3) in target blood vessels of EVT group | Immediately after the completion of endovascular therapy.
Rate of Intracranial hemorrhage (ICH) | Within 72 hours after EVT or SMT
Rate of symptomatic intracranial hemorrhage (sICH) | Within 72 hours after EVT or SMT
  The sICH was assessed based on the Heidelberg Bleeding Classification, defined as 1) ≥4 points total NIHSS at the time of diagnosis compared to immediately before worsening; 2) ≥2 point in one NIHSS category. The rationale for this is to capture new hemorrhages that produce new neurological symptoms, making them clearly symptomatic but not causing worsening in the original stroke territory; 3) Leading to intubation/hemicraniectomy/EVD placement or other major medical/surgical intervention; 4) Absence of alternative explanation for deterioration.
Rate of non-hemorrhage severe adverse event | Within 72 hours after EVT or SMT
  ulmonary infection, respiratory failure, heart failure, myocardial infarction, urinary infection, etc.
Surgical instrument-related Complications | Within 72 hours after EVT or SMT
  Vascular perforation, arterial dissection, arterial embolism, or distal embolism, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China